CLINICAL TRIAL: NCT05690386
Title: New InsiGHTS: A Multicenter, Phase 2, Randomized, Open-label, Active-controlled, Parallel Group Clinical Trial to Investigate the Safety, Tolerability, and Efficacy of Different Dose Levels of Once-weekly Lonapegsomatropin Compared to Daily Somatropin in Prepubertal Individuals With Turner Syndrome
Brief Title: A Trial to Investigate Different Doses of Lonapegsomatropin Compared to Somatropin in Individuals With Turner Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASND0034
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — lonapegsomatropin; Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: An open label, parallel group with subjects randomized into 1 of 4 treatment groups (1:1:1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lonapegsomatropin at 0.24 mg hGH/kg/week (Experimental): Lonapegsomatropin at 0.24 mg hGH/kg/week administered once-weekly by subcutaneous injection
  Interventions: Biological: Lonapegsomatropin
- Lonapegsomatropin at 0.30 mg hGH/kg/week (Experimental): Lonapegsomatropin at 0.30 mg hGH/kg/week administered once-weekly by subcutaneous injection
  Interventions: Biological: Lonapegsomatropin
- Lonapegsomatropin at 0.36 mg hGH/kg/week (Experimental): Lonapegsomatropin at 0.36 mg hGH/kg/week administered once-weekly by subcutaneous injection
  Interventions: Biological: Lonapegsomatropin
- Somatropin at 0.05 mg/kg/day (Active Comparator): Somatropin at 0.05 mg/kg/day administered once-daily by subcutaneous injection
  Interventions: Drug: Somatropin

INTERVENTIONS:
Biological: Lonapegsomatropin — Once-weekly subcutaneous injection of Lonapegsomatropin
  Arms: Lonapegsomatropin at 0.24 mg hGH/kg/week; Lonapegsomatropin at 0.30 mg hGH/kg/week; Lonapegsomatropin at 0.36 mg hGH/kg/week
Drug: Somatropin — Once-daily subcutaneous injection of Somatropin
  Arms: Somatropin at 0.05 mg/kg/day

SUMMARY:
A 104 week dose finding open label trial followed by an optional 78 week open label extension of lonapegsomatropin, a long-acting growth hormone product, administered once-a-week versus daily somatropin product in prepubertal individuals with Turner syndrome. Approximately 48 individuals (12 individuals per arm) will be randomized to receive one of three doses of lonapegsomatropin or a daily injection of somatropin. This is a trial that will be conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 and 10 years, inclusive.
2. TS diagnosis via genetic test.
3. Prepubertal status.
4. Naïve to growth hormone therapy or growth hormone secretagogue.
5. Exhibit impaired growth defined by at least one of the following:

   1. AHV< 6 cm/year or <25ᵗʰ percentile over a time span of 6-18 months for children of 2 years and older.
   2. Height (or length for individuals < 2 years old) <10ᵗʰ percentile for sex and age according to the 2000 CDC Growth Charts for the United States.
6. Bone age within normal limits for chronological age, defined as no more than 20% above or below chronological age in months or delayed for chronological age (greater than 20% below chronological age), at screening.
7. Biochemically euthyroid (including when on thyroid hormone supplementation).
8. If on hormone replacement therapies for any hormone deficiencies other than growth hormone (e.g. adrenal, thyroid), must be on adequate and stable doses for ≥4 weeks prior to and throughout Screening.
9. Fundoscopy at Screening without signs/symptoms of intracranial hypertension or proliferative retinopathy or evidence of any other retinal disease for which growth hormone therapy is contraindicated.
10. Capable of giving signed informed consent. Participants and/or parents or legal guardians of participants must sign an informed consent statement. Assent should be obtained from all participants competent to understand the protocol, per IRB requirements.

Exclusion Criteria:

1. Turner Syndrome with presence of Y-chromosomal material on genetic testing and without a history of gonadectomy.
2. Diagnosis of diabetes mellitus.
3. Known history of clinically relevant conditions that may have an effect on growth, e.g. but not limited to celiac disease, malnutrition, treatment with potential growth-influencing medications for Attention-deficit/ hyperactivity disorder (ADHD), etc.
4. Any known, clinically significant, congenital or acquired cardiac/cardiovascular dysfunction that might interfere with growth as determined by transthoracic echocardiogram.
5. Known history or presence of malignancy.
6. Individuals with history of intracranial tumor or cysts, with evidence of growth within the last 12 months prior to Screening.

   Note - Individuals with a history of intracranial tumor may be eligible if there is no evidence of residual tumor as determined by MRI/CT scan(s) performed within 6 to 12 months prior to screening.
7. Hepatic transaminases (i.e., AST or ALT) above 3 times the upper limit of normal according to the central laboratory at screening.
8. Major medical conditions and/or presence of contraindication to hGH treatment.
9. Abnormal renal function.
10. Clinically relevant systemic illness, acute critical illness, and complications following open heart surgery, abdominal surgery, multiple accidental traumas, acute respiratory failure, or similar conditions within 6 months prior to Screening.
11. Poorly controlled hypertension.
12. Receiving prior or concurrent treatment with any agent that might influence growth or interfere with GH secretion or action such as, but not limited to, non steroidal anabolic agents, sex steroids, etc.
13. Oral/intravenous/intramuscular corticosteroids within 90 days prior to or throughout Screening.
14. Known or suspected hypersensitivity to study intervention(s) or related products.
15. Participation in any other trial involving an investigational compound within 90 days prior to Screening or in parallel to this trial.
16. Any disease or condition that, in the judgement of the investigator, may make the individual unlikely to comply with the protocol or presents undue risk.
17. Female who is pregnant, plans to be pregnant, or is breastfeeding.

Ages: 1 Year to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Annualized Height Velocity (AHV) (cm/year) | 26 weeks
  Calculated based on the difference between the AHV at 6 months and baseline

SECONDARY OUTCOMES:
Annualized Height Velocity (AHV) (cm/year) | 52 weeks, 104 weeks, 156 weeks and 182 weeks
  Calculated based on the difference between the AHVs at 12, 24, 36 and 42 months and baseline
Change from baseline in height standard deviation score (SDS) | 26 weeks, 52 weeks, 104 weeks, 156 weeks and 182 weeks
  Calculated based on the difference between the heights SDS at 6, 12, 24, 36 and 42 months and baseline
Change from baseline in Bone age (calculated years) | 52 weeks, 104 weeks and 156 weeks
  Annual change in bone age measurements as per Gruelich-Pyle method
Change from baseline in ratio of bone age/chronological age | 52 weeks, 104 weeks and 156 weeks
  Calculated as a ratio

OTHER OUTCOMES:
Insulin-like growth factor 1 (IGF-1) standard deviation score (SDS) | 26 weeks, 52 weeks, 104 weeks, 156 weeks and 182 weeks
  Via Central Lab analysis

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Ascendis Pharma Investigational Site, Palo Alto, California
  - Ascendis Pharma Investigational Site, San Diego, California
  - Ascendis Pharma Investigational Site, Aurora, Colorado
  - Ascendis Pharma Investigational Site, Orlando, Florida
  - Ascendis Pharma Investigational Site, St. Petersburg, Florida
  - Ascendis Pharma Investigational Site, Atlanta, Georgia
  - Ascendis Pharma Investigational Site, Idaho Falls, Idaho
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Boston, Massachusetts
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Las Vegas, Nevada
  - Ascendis Pharma Investigational Site, Lake Success, New York
  - Ascendis Pharma Investigational Site, Chapel Hill, North Carolina
  - Ascendis Pharma Investigational Site, Cincinnati, Ohio
  - Ascendis Pharma Investigational Site, Oklahoma City, Oklahoma
  - Ascendis Pharma Investigational Site, Portland, Oregon
  - Ascendis Pharma Investigational Site, El Paso, Texas
  - Ascendis Pharma Investigational Site, Fort Worth, Texas
  - Ascendis Pharma Investigational Site, Seattle, Washington